CLINICAL TRIAL: NCT01536821
Title: PROGENI (Parkinson's Research: The Organized Genetics Initiative) Family Study
Brief Title: PROGENI (Parkinson's Research: The Organized Genetics Initiative) Family Study of LRRK2 (Leucine-rich Repeat Kinase 2)
Acronym: PROGENI
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: 1105005340
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Parkinson's Disease; PD; LRRK2; genetics; genes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma and serum will be obtained and stored from a blood sample. In addition, a whole blood and urine samples will be obtained and stored.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The PROGENI Family Study is part of a larger consortium that is studying a gene shown to be important in Parkinson's disease, called LRRK2. People who have a defect in the LRRK2 gene will often develop Parkinson's disease. Eligible participants will be asked to complete a single Study Visit at an affiliated research facility closest to their home.

DETAILED DESCRIPTION:
Participants will be asked to complete a family history questionnaire, which will gather information about their family history of Parkinson's disease and related disorders. They will be asked to complete a single Study Visit, during which they will be asked to do some or all of the following:

1. Complete questionnaires regarding Parkinson's disease symptoms, medical history, mood, sleep, mental status, and activity level.
2. Be given a brief standard neurological examination.
3. Be given a scratch and sniff smell identification test.
4. Be asked to give a sample of approximately 2 tablespoons of blood.
5. Be asked to give a urine sample of approximately 1 tablespoon of urine.

ELIGIBILITY:
Inclusion Criteria:

Positive for a LRRK2 mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must provide test results documenting a LRRK2 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Observation and biological specimen collection | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Foroud, PhD, Principal Investigator — Indiana University
Locations (10):
- United States (9):
  - Cleveland Clinic Florida, Weston, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Nebraska, Omaha, Nebraska
  - Beth Israel Medical Center, New York, New York
  - Medical University of Ohio, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
- University of Alberta, Edmonton, Alberta, Canada